CLINICAL TRIAL: NCT02901587
Title: Interventional, Randomised, Double-blind, Parallel-group, Active-control, Multiple-dose Study Investigating the Effect of Lu AF35700 on Cardiac Repolarization in Men and Women With Schizophrenia and Schizoaffective Disorder
Brief Title: Study Investigating the Effect of Lu AF35700 on Cardiac Repolarization in Men and Women With Schizophrenia and Schizoaffective Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16323A
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Lu AF35700; Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lu AF35700 (10 mg/day) (Experimental): Lu AF35700 10 mg/day for 6 weeks
  Interventions: Drug: Lu AF35700 (10 mg/day)
- Lu AF35700 (30 mg/day) (Experimental): Lu AF35700 30 mg/day for 6 weeks
  Interventions: Drug: Lu AF35700 (30 mg/day)
- Quetiapine (Seroquel XR® 800 mg/day) (Experimental): Quetiapine (Seroquel XR®) 800 mg/day for 6 weeks
  Interventions: Drug: Quetiapine (Seroquel XR® 800 mg/day)

INTERVENTIONS:
Drug: Lu AF35700 (10 mg/day) — tablets for oral administration once daily
  Arms: Lu AF35700 (10 mg/day)
Drug: Lu AF35700 (30 mg/day) — tablets for oral administration once daily
  Arms: Lu AF35700 (30 mg/day)
Drug: Quetiapine (Seroquel XR® 800 mg/day) — tablets for oral administration once daily
  Arms: Quetiapine (Seroquel XR® 800 mg/day)

SUMMARY:
The purpose of this study is to investigate the effect of Lu AF35700 on electrical activity in the heart as measured on an electrocardiogram (ECG) in patients with schizophrenia or schizoaffective disorder after 6 weeks of treatment

ELIGIBILITY:
Inclusion Criteria:

* The patient is able by her/himself to provide informed consent to participate in the study
* The patient has a primary diagnosis of schizophrenia or schizoaffective disorder (DSM-5™ criteria)
* The patient has BMI ≤35 kg/m2
* The patient has a Clinical Global Impression - Severity of Illness (CGI-S) score ≤4 (moderately ill)
* PANSS total score ≤ 80 and a score ≤4 (moderate) on the PANSS items, P7 (hostility) and G8 (uncooperativeness)
* The patient is willing to be hospitalized for up to 8 weeks
* The patient is generally healthy based on medical history, physical examination, vital signs, ECG, and laboratory tests.
* The patient agrees to protocol-defined use of effective contraception

Exclusion Criteria:´

* The patient experienced acute exacerbation of psychosis requiring hospitalization within the last 3 months or required change in medication due to exacerbation of psychosis within the last 8 weeks
* The patient has met moderate or severe co-morbid Substance Abuse Disorder DSM-5™ criteria in the last 3 months
* The patient is at significant risk of harming her/himself or others in the opinion of the investigator or according to Columbia Suicide Severity Rating Scale (C-SSRS)
* The patient has tested positive for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (anti-HCV)

Other protocol defined inclusion and exclusion criteria may apply

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
Change from time-matched baseline on day 1, 21, and 42 in QTcF | Before dose to 10 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- US1104, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No